CLINICAL TRIAL: NCT00358904
Title: Assessment of Weber Humeral Derotational Osteotomy Using CT Scan
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. William Regan, University of British Columbia
Other Study IDs: C05-0678
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-04

CONDITIONS: Hill Sachs
Keywords: Hill Sachs; Weber osteotomy; shoulder dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Subjects who have had the Weber osteotomy for Hill-Sachs lesions will have CT of Both shoulders. Amount of rotation in operative shoulder will be compared to contralateral. QOL will be assessed

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have had the Weber osteotomy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have had the Weber osteotomy for Hill-Sachs lesions.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2006-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Regan, MD, Principal Investigator — The University of British Columbia
Locations (1):
- Vancouver General Hospital, Orthopaedics Dept., Vancouver, British Columbia, Canada